CLINICAL TRIAL: NCT07383818
Title: A Prospective, Multigroup, Multi-center, Open-label Clinical Study of Trastuzumab Rezetecan as Neoadjuvant Therapy Combined With Toripalimab in HR+/HER2-low Breast Cancer Patients (NEOTORCH-BREAST 08)
Brief Title: Neoadjuvant Therapy Combined With Trastuzumab Rezetecan and Toripalimab for HR+/HER2-low Breast Cancer (NEOTORCH-BREAST 08)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250148C-R1
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: HR Positive/HER2 Low Breast Cancer
Keywords: Breast cancer; Toripalimab; Trastuzumab Rezetecan; Neoadjuvant therapy; HR Positive/HER2 Low Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — toripalimab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neoadjuvant therapy combined with Trastuzumab Rezetecan and Toripalimab (Experimental): Drug: Neoadjuvant therapy combined with Trastuzumab Rezetecan and Toripalimab Description:Trastuzumab Rezetecan administered intravenously at a dose of 4.8mg/kg every 3 weeks for a total of 24 weeks with Toripalimab intravenous infusion of 240mg. During postoperative adjuvant therapy, Toripalimab used as before till a total of 1 year.
  Interventions: Drug: Neoadjuvant therapy combined with Trastuzumab Rezetecan and Toripalimab
- Neoadjuvant chemotherapy combined Toripalimab (Experimental): Drug: Neoadjuvant Chemotherapy in Combination with Toripalimab Description: Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks. During neoadjuvant chemotherapy and postoperative adjuvant therapy, use of Toripalimab: intravenous infusion of 240 mg, once every 3 weeks, combined with preoperative neoadjuvant and postoperative adjuvant therapy for a total of 1 year.
  Interventions: Drug: Neoadjuvant Chemotherapy in Combination with Toripalimab
- Neoadjuvant Chemotherapy (Other): Drug: Neoadjuvant Chemotherapy Description: Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks.
  Interventions: Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant therapy combined with Trastuzumab Rezetecan and Toripalimab — Trastuzumab Rezetecan administered intravenously at a dose of 4.8mg/kg every 3 weeks for a total of 24 weeks with Toripalimab intravenous infusion of 240mg. During postoperative adjuvant therapy, Toripalimab used as before till a total of 1 year.
  Arms: Neoadjuvant therapy combined with Trastuzumab Rezetecan and Toripalimab
Drug: Neoadjuvant Chemotherapy in Combination with Toripalimab — Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks. During neoadjuvant chemotherapy and postoperative adjuvant therapy, use of Toripalimab: intravenous infusion of 240 mg, once every 3 weeks, combined with preoperative neoadjuvant and postoperative adjuvant therapy for a total of 1 year.
  Arms: Neoadjuvant chemotherapy combined Toripalimab
Drug: Neoadjuvant Chemotherapy — Epirubicin (or Liposomal Doxorubicin)+Cyclophosphamide, intravenous infusion of 100 mg/m2. Epirubicin (or 35 mg/m2 liposomal doxorubicin)+600 mg/m2 cyclophosphamide, starting from the first day of the week, for a total of 12 weeks. Paclitaxel, administered intravenously at a dose of 260 mg/m2 every 3 weeks for a total of 12 weeks.
  Arms: Neoadjuvant Chemotherapy

SUMMARY:
This study is a prospective, multi-cohort, multicenter, open-label exploratory clinical trial. The primary study objective is to evaluate the pathologic complete response (PCR) of treatment of HR+/HER2-low breast cancer with neoadjuvant therapy combined with Trastuzumab Rezetecan and Toripalimab , including the incidences and types of adverse events. The secondary endpoints include event-free survival (EFS), residual cancer burden (RCB), and objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years old;
2. ECOG score is 0-1 points;
3. Histologically or pathologically confirmed invasive breast cancer, meeting the following criteria simultaneously: Invasive breast cancer staged as T1cN1-2M0 or T2-3N0-2M0; All patients must be pathohistologically confirmed as HR-positive/HER2-low. The interpretation of ER and PR status follows the 2020 ASCO/CAP Guidelines: expression ≥1% is defined as positive, and HR positivity is confirmed if either ER or PR is positive. The interpretation of HER2 status follows the 2023 ASCO/CAP Guidelines: HER2-low is defined as HER2 1+ or 2+ with negative FISH test results. Pathological testing for PD-L1 expression: The Combined Positive Score (CPS) is the percentage of PD-L1-positive cells (including tumor cells, lymphocytes, and macrophages) among the total number of tumor cells. The PD-L1 antibody clone used for detection at our center is 22C3. No prior anti-cancer treatment.
4. Function levels of major organs must meet the required criteria
5. For female patients who have not yet reached menopause or undergone surgical sterilization: during the treatment period and in the study treatment, the final use effective contraceptive methods for at least 6 months after a single administration.
6. Voluntarily join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Stage IV breast cancer.
2. Inflammatory breast cancer.
3. Previously received anti-tumor treatment or radiation therapy for any malignant tumor, excluding those that have been cured Malignant tumors such as cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma.
4. Simultaneously undergoing anti-tumor treatment in other clinical trials, including but not limited to chemotherapy and endocrine therapy. Treatment, biological therapy, bone improvement drug therapy, or immune checkpoint inhibitor therapy, etc.
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before the first administration of the study drug, or the patient has not fully recovered from such surgical procedures.
6. Serious heart disease or discomfort.
7. Uncontrolled active infections that require treatment; History of immunodeficiency, including HIV testing positive Sexual, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.
8. Patients with chronic active hepatitis B or active hepatitis C
9. Have received immunotherapy and experienced adverse immune events such as immune related pneumonia and myocarditis, which have been determined by researchers to potentially affect the safety of the experimental medication.
10. Individuals with a known history of allergies to the components of this medication regimen.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（PCR） | 2 years

SECONDARY OUTCOMES:
Event free survival (EFS) | 5 years
objective response rate (ORR) | 5 years
Residual Cancer Burden (RCB) | 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Zhongshan Hospital, Fudan University, Shanghai
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No